CLINICAL TRIAL: NCT00026897
Title: Trafficking of Indium-111-Labeled Cultured Immune Cells in Patients Undergoing Immunotherapy for Advanced Cancer
Brief Title: Trafficking of Indium-III-Labeled Cultured Immune Cells in Patients Undergoing Immunotherapy for Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980033; 98-C-0033
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-12

CONDITIONS: Neoplasm
Keywords: Adoptive Immunotherapy; Cellular Therapy; Lymphocyte Migration; Tumor Imaging
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Procedure: Gamma-camera imaging
Procedure: Low-risk biopsy

SUMMARY:
Patients undergoing immunotherapy for advanced cancer under IRB-approved protocols, who are to receive immune cells in adoptive transfer, will have less than or equal to 50% of those cells labeled with In-111-oxine and administered along with the remainder of their unlabeled cells. They will then undergo gamma-camera imaging over the next 0-7 days and blood samples and tumor sites which are accessible with minimal surgery (low-risk biopsy) may be sampled in some patients for enumeration of radiolabeled cells. End-points will be tumor and normal organ imaging and the amount of In-111 per gram of tissue in biopsies or per ml. of blood.

DETAILED DESCRIPTION:
Patients undergoing immunotherapy for advanced cancer under IRB-approved protocols, who are to receive immune cells in adoptive transfer, will have less than or equal to 50% of those cells labeled with In-111-oxine and administered along with the remainder of their unlabeled cells. They will then undergo gamma-camera imaging over the next 0-7 days and blood samples and tumor sites which are accessible with minimal surgery (low-risk biopsy) may be sampled in some patients for enumeration of radiolabeled cells. End-points will be tumor and normal organ imaging and the amount of In-111 per gram of tissue in biopsies or per ml. of blood.

ELIGIBILITY:
INCLUSION CRITERIA

All patients will be 18 years of age or older.

All patients will be enrolled in NCI-approved intramural immunotherapy protocol in which immune cells are adoptively administered to treat advanced cancer.

EXCLUSION CRITERIA

Patients who are receiving less than 3x10(9) cells in transfer will be excluded.

Impaired patients who are unable to give valid informed consent will also be excluded.

Patients who are pregnant will be excluded.

All other exclusion criteria stated in the parent immunotherapy protocol.

Patients who are HIV-infected.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1997-12; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Shu S, Chou T, Rosenberg SA. In vitro sensitization and expansion with viable tumor cells and interleukin 2 in the generation of specific therapeutic effector cells. J Immunol. 1986 May 15;136(10):3891-8. PMID 3486223
- [Background] Shu SY, Chou T, Rosenberg SA. Generation from tumor-bearing mice of lymphocytes with in vivo therapeutic efficacy. J Immunol. 1987 Jul 1;139(1):295-304. PMID 2953816
- [Background] Rosenberg SA, Packard BS, Aebersold PM, Solomon D, Topalian SL, Toy ST, Simon P, Lotze MT, Yang JC, Seipp CA, et al. Use of tumor-infiltrating lymphocytes and interleukin-2 in the immunotherapy of patients with metastatic melanoma. A preliminary report. N Engl J Med. 1988 Dec 22;319(25):1676-80. doi: 10.1056/NEJM198812223192527. PMID 3264384